CLINICAL TRIAL: NCT04718948
Title: "The Feasibility of a Multimodal Spectroscopy Analysis to Detect Urothelial Cancer in Urine"
Brief Title: Multimodal Spectroscopy to Detect Urothelial Cancer in Urine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Florence (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); European Laboratory for Non-Linear Spectroscopy (Unknown); Careggi Hospital (Other)
Responsible Party: Principal Investigator, Simone Morselli, MD, University of Florence
Other Study IDs: 17686_BIO
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Urothelial Carcinoma; Urinary Bladder Cancer; Urinary Tract Cancer
Keywords: Urinary Tract Cancer; Urine; Spectroscopy; Laser; Urine Cytology
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Urologic Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients Positive for Urinary Tract Cancer: Patients will undergo urinary cytology, multimodal spectroscopy in urine and urologic surgical intervention
  The group of cases will consist of patients who meet the inclusion and exclusion criteria in the operative note for:
  * Transurethral Resection of Bladder Neoplasia (TURBT)
  * Radical Cystectomy for Bladder Neoplasia
  * Diagnostic ureterorenoscopy and / or laser treatment of ureteral and / or renal pelvis neoplasia
  * Segmental ureterectomy with or without ureteral reimplantation
  * Nephroureterectomy with or without bladder cuff excission
  Interventions: Device: Urinary Multimodal Fiber Optic Spectroscopy; Diagnostic Test: Urine Cytology; Procedure: Surgery
- Patients Negative for Urinary Tract Cancer: Patients will undergo urinary cytology, multimodal spectroscopy in urine and urologic surgical intervention
  The control group will consist of patients who meet the inclusion and exclusion criteria in the operative note for:
  * Transurethral Resection of Prostate (TURP)
  * Other endoscopic treatments of Benign Prostatic Hyperplasia (BPH)
  * Open interventions of prostatic adenomectomy
  * Endoscopic lithotripsy interventions of bladder stones or cystotomy with removal of bladder stones
  * Rigid and / or flexible ureterorenoscopy for the treatment of kidney and / or ureteral stones
  * Placement of ureteral catheter for ureteral and / or renal stones
  * Bladder Neck Incision (TUIP)
  * Endoscopic urethrotomy
  Interventions: Device: Urinary Multimodal Fiber Optic Spectroscopy; Diagnostic Test: Urine Cytology; Procedure: Surgery

INTERVENTIONS:
Device: Urinary Multimodal Fiber Optic Spectroscopy — Approach based on a physical principle, mainly spectroscopy, which is rapid non-invasive and does not require the use of additional substances or contrast media in the diagnosis of urothelial neoplasms in urine samples.
  It will be administered through a appositely designed device
Diagnostic Test: Urine Cytology — An expert cytopathologist will analyze urine samples to detect urinary tract cancer cells. It is the current golden standard to detect urothelial cancer in urine
Procedure: Surgery — It will provide a reliable information on the presence/absence of cancer in the urinary tract (from direct visualization to pathological analysis)

SUMMARY:
To facilitate the follow-up of urothelial tumors and also make them more tolerable and less invasive for patients, there is a minimally invasive and easy to perform examination which is urinary cytology on 3 samples. This test is extremely specific, over 90% chance of cancer if it is positive and is performed by expert cytopathologists, but it is burdened by a very low sensitivity, which is especially acute in the case of low grade tumors. This makes it an extremely useful test in case of positivity, but of little use if negative or doubtful, not being able to consider it reliable.

To overcome this problem, our study aims to bring an approach based on a physical principle, that is spectroscopy, which is fast non-invasive and does not require the use of additional substances or contrast media in the diagnosis of urothelial neoplasms in samples of urine.

In our experience, multimodal optical fiber spectroscopy has proved extremely valid in discriminating healthy urothelial tissue from tumor ex vivo, as well as providing important information on the degree of urothelial neoplasia, with accuracy rates higher than 80%, for which developed the idea of a technique based on multimodal spectroscopy.

If our method proves valid, it could improve the follow up and management of patients with urothelial cancer, being able to support normal cytology and provide further support to the cytopathologist, as well as simplify the diagnosis.

ELIGIBILITY:
CASES Inclusion criteria

Patients over the age of 18 who are known for urological interventions for the following pathologies will be considered for enrollment in the group of cases:

* Bladder cancer
* Urethral tumor
* Renal Pelvis Tumor
* Ureteral tumor

The exclusion criteria will be:

* Age under 18
* Pregnancy
* Lack of informed consent
* Persons with indwelling catheter
* Presence of prostate cancer
* Presence and / or history of renal cancer, except tumors of the renal pelvis

CHECKS Inclusion criteria

Patients over the age of 18 who are known for urological interventions for the following pathologies will be considered for enrollment in the control group:

* Kidney, ureteral or bladder stones
* BPH

The exclusion criteria will be:

* Age under 18
* Pregnancy
* Lack of informed consent
* Indwelling Catheter wearers
* Presence of prostate cancer
* Presence of kidney cancer, including kidney pelvic tumors
* Presence and / or history of ureteral cancer
* Presence and / or history of bladder cancer
* Presence and / or history of urethral cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the inclusion and exclusion criteria will be enrolled at Urology ward admission. Informed consent will be collected. Patients therapeutic routine will be unaffected.
  In the morning before surgery, the patient will collect urine sample. The patient will then continue the previously established diagnostic therapeutic process. The sample will be brought to the spectroscopic and cytological analysis. Samples will not be stored.
  According to the sample size calculation based on the asymptotic normal distribution theory, a total of 240 cases and 240 controls will be required if the study is to have 90% power. A series of 5000 simulations generating binary test data with a true positive frequency and a true negative frequency of 80% showed that these sample sizes produce 89% power. Increasing the sample size to 250 cases and 250 controls increases the potency to 90%. Therefore, approximately 250 cases and 250 controls will be enrolled in this phase 2 validation study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-01-25 (Estimated)

PRIMARY OUTCOMES:
Urine Multimodal Spectroscopy Reliability | Enrollment
  Evaluate whether multimodal spectroscopy can discriminate between healthy controls and patients with urothelial neoplasia on urine, with an accuracy at least comparable to urinary cytology on 3 samples

SECONDARY OUTCOMES:
Urine Multimodal Spectroscopy Grading | Enrollment
  Evaluate whether multimodal spectroscopy is able to discriminate between high or low grade urothelial lesions on urine
Urine Multimodal Spectroscopy Site Discrimination | Enrollment
  Evaluate whether multimodal spectroscopy is able to discriminate between lower or upper urinary tract lesions on urine

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Gacci, MD, Principal Investigator — Careggi University Hospital; Enrico Baria, PhD, Principal Investigator — European Laboratory for Non-Linear Spectroscopy; Riccardo Cicchi, PhD, Principal Investigator — Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy; Francesco Saverio Pavone, Prof, Principal Investigator — University of Florence; Sergio Serni, Prof, Principal Investigator — University of Florence; Gabriella Nesi, Prof, Principal Investigator — University of Florence
Locations (1):
- Careggi Hospital, Florence, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baria E, Morselli S, Anand S, Fantechi R, Nesi G, Gacci M, Carini M, Serni S, Cicchi R, Pavone FS. Label-free grading and staging of urothelial carcinoma through multimodal fibre-probe spectroscopy. J Biophotonics. 2019 Nov;12(11):e201900087. doi: 10.1002/jbio.201900087. Epub 2019 Aug 13. PMID 31343832